CLINICAL TRIAL: NCT00430755
Title: Quality Assessment for History Taking With or Without an Knowledge Based Interview System.
Brief Title: Improving the Quality of Patient Care by Using a Clinical Expert System.
Acronym: CLEOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Responsible Party: Principal Investigator, Dominik M. Alscher, MD, Chief Medical Officer, Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RBK080
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension; Diabetes; Hypercholesterolemia; Vasculitis; Coronary Heart Diseases
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Hypercholesterolemia; Vasculitis; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inpatients of hospital (Other): All patients who were admitted to the departments of nephrology or cardiology in a tertiary hospital in Germany.
  The intervention was use of an expert system to acquire medical histories by direct interview of patients.
  Description of the software program - The program tested in this study consisted of a data acquisition [history-taking] component and a data analysis component. The data acquisition component was constructed on the basis of established principles of pathophysiology. Medical knowledge was formalized as software algorithms that were machine-readable by representing the knowledge as branched chain decision trees.
  Interventions: Device: Computer-assisted history; Procedure: physician taken history; Other: Computer-assisted history taking

INTERVENTIONS:
Device: Computer-assisted history — Methods The intervention was use of an expert system to acquire medical histories by direct interview of patients.
  Description of the software program - The program tested in this study consisted of a data acquisition [history-taking] component and a data analysis component. The data acquisition component was constructed on the basis of established principles of pathophysiology. Medical knowledge was formalized as software algorithms that were machine-readable by representing the knowledge as branched chain decision trees.
  Other Names: CLEOS
Procedure: physician taken history — Convential history taking by physicians
  Other Names: Traditional history taking
Other: Computer-assisted history taking

SUMMARY:
Aim:

To investigate the quality of history taking by physician and computer-based system.

Patients:

100 inpatients presenting at the RBK for the first time and treated in the departments of nephrology and cardiology.

Methods:

The information obtained by the computer based system is compared with the information acquired by conventional history taking. Study endpoint is the comparison of historical data organized according to the elements in a standard medical history on a patient-by-patient basis.

Study procedure History taking is performed by physicians according to the guidelines of the RBK. Within 2 days thereafter the patient is interviewed with help of the CLEOS system with the support of a study nurse.

DETAILED DESCRIPTION:
Aim:

To compare the completeness of history taking by physicians and by a computerized system interacting directly with the patients. Historical data recorded in the patient record, including the discharge letter, were compared with the history acquired by computer-based interview of each patient.

Patients:

100 inpatients presenting at the RBK for the first time and treated in the departments of nephrology and cardiology.

Methods:

The information obtained by the computer based system is compared with the information acquired by conventional history taking. Study endpoint is the comparison of historical data organized according to the elements in a standard medical history on a patient-by-patient basis.

Study procedure After informed consent of the patients the procedure of history taking is performed by the physician according to the guidelines of the RBK. Within 2 days thereafter the patient is interviewed with help of the CLEOS system [a computer-based, history-taking program] with the support of a study nurse. The physician will be informed about the results immediately after completion of the questionnaire.

Data of medical significance were extracted from the official hospital chart and the computerized history by clinically experienced physicians and tabulated on a patient-by-patient basis. data elements were compared across each category of the history for each patient interviewed. The relevance of the differences of the information obtained by the two systems was rated by an independent reviewer.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients in a hospital environment

Exclusion Criteria:

* Inability to give an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2005-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominik M Alscher, MD, Principal Investigator — Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Locations (1):
- Robert-Bosch-Hospital, Stuttgart, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were interviewed had been admitted emergently. Patient charts were not consulted prior to any interview; and the study nurse, who picked patients randomly for interview, had no knowledge of these patients before an interview and carried on no discussions with floor staff about a patient's clinical state.
Pre-assignment Details: Acquisition of clinical data in the history-taking program is based on the principles of pathophysiology formalized as software algorithms representing medical knowledge as branched chain decision trees.
Groups:
- Inpatients With the Need for History Taking: Every patient, who needs to get a medical history taken
Period: Overall Study
Arm/Group | Inpatients With the Need for History Taking
Started | 98
Completed | 45
Not Completed | 53
Not completed — Withdrawal by Subject | 53

BASELINE CHARACTERISTICS:
Arm/Group | Inpatients With the Need for History Taking
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 57
Region of Enrollment [Number; unit: participants]
  Germany | 98

OUTCOME MEASURES:

1. Primary Outcome: Detection of Medical Problems (by Number of Problems Reported by Computer Assisted History, That Were Not Reported by Physician Taken History)
Description: Data were extracted from hospital charts by to experienced physicians.; data from the computer histories were extracted by a senior physician, who tabulated comparisons between the 2 sets of records. We used the number of problems reported by Computer Assisted History that were not reported by Physician. Nurses at Robert Bosch Krankenhaus do not take medical histories in regard to allergies or adverse drug reactions. Pharmacists make no entries into charts and have no separate records of drug allergies or history of adverse drug reactions. Data on these issues either are obtained only by physician interview of the patient.
Time Frame: participants were followed for the duration of hospital stay, an average of 8 days
Population: The rest did not end the history tool
Measure: Number; unit: medical problems
Arm/Group | Inpatients With the Need for History Taking
Number analyzed (Participants) | 98
medical problems | 98

ADVERSE EVENTS:
Arm/Group | Inpatients With the Need for History Taking
Serious Adverse Events (participants affected / at risk) | 0/98
Other Adverse Events (participants affected / at risk) | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes